CLINICAL TRIAL: NCT01898923
Title: Randomized Controlled Study to Evaluate the Efficacy and Safety of ON101 Cream for the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Evaluate the Efficacy and Safety of ON101 Cream for the Treatment of Chronic Diabetic Foot Ulcers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ON101CLCT02
Record Dates: First submitted 2013-07-08; First posted 2013-07-15 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-03

CONDITIONS: Diabetic Foot
Keywords: WH-1,Diabetic Foot,Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ON101 Cream (Experimental): ON101 Cream (1.25%),15g ointment per tube. Twice daily for up to 16 weeks.
  Interventions: Drug: ON101 Cream
- Aquacel® Hydrofiber® dressing (Other): Aquacel® Hydrofiber® dressings will be changed daily, on alternate days or three times a week according to need, but not longer than 7 days.
  Interventions: Other: Aquacel® Hydrofiber® dressing

INTERVENTIONS:
Drug: ON101 Cream
  Other Names: WH-1
  Arms: ON101 Cream
Other: Aquacel® Hydrofiber® dressing
  Arms: Aquacel® Hydrofiber® dressing

SUMMARY:
The primary objective of this study is to evaluate the efficacy of the new treatment of WH-1 ointment compared to Aquacel® Hydrofiber® dressing, applied to chronic diabetic foot ulcers for up to 16 weeks.An additional objective of this study is to collect safety information including adverse events and clinical laboratory abnormalities.

DETAILED DESCRIPTION:
This trial is designed as a randomized, evaluator blinded, active-controlled, multi-center study comparing the efficacy and safety of WH-1 ointment and Aquacel® Hydrofiber® dressing in the treatment of diabetic foot ulcers. Independent evaluators who blinded to subjects' treatment will evaluate whether the wound has healed. Eligible subjects will be randomized to receive either WH-1 ointment or Aquacel® Hydrofiber® dressing in a 1:1 allocation. The study treatment will be applied to the selected ulcer for a maximum period of 16 weeks, until the wound/ulcer closure (wound size of 0) for two consecutive visits at least 2 weeks apart, or until the subject exited the study as treatment failure. After that, all subjects regardless of wound healing at the end of comparison period will be followed for 12 weeks to investigate durability. During the follow-up period, Aquacel® Hydrofiber® dressing will be applied for subjects who have unhealed or with recurrent wound. Each target ulcer with wound photographs for blind assessment will be monitored at each scheduled visit.

One interim analysis is planned at around 50% of study information; the final analysis will be conducted at the end of the study.

ELIGIBILITY:
Inclusion Criteria

1. Has signed a written informed consent prior to the first study evaluation;
2. Male or female is at least 20 and < 80 years of age;
3. Diabetes mellitus (type 1 or 2) with an HbA1c < 12.0% measured during screening or within three months prior to randomization;
4. An ankle brachial index on the target limb at least 0.8 measured during screening or within three months prior to randomization;
5. The target ulcer must have the following characteristics:

   * Grade 1 or 2 per Wagner Ulcer Classification System;
   * No higher than the ankle;
   * No active infected;
   * A cross-sectional area of between 1 and 25 cm2 post-debridement;
   * Present for at least 4 weeks before randomization;
6. If female and of childbearing potential has a negative pregnancy test and is not breastfeeding at screening visit;
7. Able and willing to attend the scheduled visits and comply with study procedures.

Exclusion Criteria:

1. Presence of necrosis, purulence or sinus tracts that cannot be removed by debridement;
2. Acute Charcot's neuroarthropathy as determined by clinical and/or radiographic examination;
3. Has undergone revascularization procedure aimed at increasing blood flow in the treatment target limb < 4 weeks prior to randomization;
4. Poor nutritional status defined as an albumin < 2.5 g/dL;
5. Aspartate Aminotransferase(AST, GOT) and/or Alanine Aminotransferase(ALT, GPT) >3 x the normal upper limit;
6. Serum Creatinine >2 x the normal upper limit;
7. Treatment with immunosuppressive or chemotherapeutic agents, radiotherapy or systemic corticosteroids less than 4 weeks before randomization;
8. Use of any investigational drug or therapy within the 4 weeks prior to randomization;
9. A psychiatric condition (e.g., suicidal ideation), current or chronic alcohol or drug abuse problem, determined from the subject's medical history, which, in the opinion of the Investigator, may pose a threat to subject compliance;
10. Judged by the investigator not to be suitable for the study for any other reason.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2012-11-23 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Chang, Study Director — Oneness Biotech
Locations (21):
- Limb Preservation Platform, Inc., Fresno, California, United States
- China (9):
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guanzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guanzhou, Guangdong
  - The First Affiliated Hospital of Henan Science & Technology University, Luoyang, Henan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Shandong Provincial Hospital, Jinan, Shandong
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai TCM-Interated Hospital, Shanghai, Shanghai Municipality
- Taiwan (11):
  - Chang Gung Medical Hospital_Kaohsiung, Kaohsiung City
  - Buddhist Tzu Chi Medical Hospital, New Taipei City
  - MacKay Memorial Hospital-Tamsui Branch, New Taipei City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center-Yongkang, Tainan
  - MacKay Memorial Hospital-Taipei Branch, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Medical Hospital_Linkou, Taoyuan
  - China Medical University Hospital-Beigang Branch, Yunlin

REFERENCES:
- [Derived] Huang YY, Lin CW, Cheng NC, Cazzell SM, Chen HH, Huang KF, Tung KY, Huang HL, Lin PY, Perng CK, Shi B, Liu C, Ma Y, Cao Y, Li Y, Xue Y, Yan L, Li Q, Ning G, Chang SC. Effect of a Novel Macrophage-Regulating Drug on Wound Healing in Patients With Diabetic Foot Ulcers: A Randomized Clinical Trial. JAMA Netw Open. 2021 Sep 1;4(9):e2122607. doi: 10.1001/jamanetworkopen.2021.22607. PMID 34477854

RESULTS

PARTICIPANT FLOW:
Groups:
- ON101 Cream: ON101 Cream (1.25%),15g ointment per tube. Twice daily for up to 16 weeks.
  ON101 Cream
- Aquacel® Hydrofiber® Dressing: Aquacel® Hydrofiber® dressings will be changed daily, on alternate days or three times a week according to need, but not longer than 7 days.
  Aquacel® Hydrofiber® dressing
Period: Overall Study
Arm/Group | ON101 Cream | Aquacel® Hydrofiber® Dressing
Started | 122 | 114
Completed | 106 | 93
Not Completed | 16 | 21
Not completed — Lack of Efficacy | 5 | 6
Not completed — Adverse Event | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 4 | 7
Not completed — Physician Decision | 3 | 4
Not completed — One of the subjects IS NO LONGER USING AQUACEL STANDARD OF CARE AND WAS REMOVED FROM THE STUDY | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ON101 Cream | Aquacel® Hydrofiber® Dressing | Total
Number analyzed (Participants) | 122 | 114 | 236
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (10.6) | 56.6 (11.3) | 57.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 32 | 61
  Male | 93 | 82 | 175
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
  China | 20 | 20 | 40
  Taiwan | 98 | 90 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Ulcer Closure
Description: The primary variable is the number of target ulcers healed in each group within 16 weeks. The primary efficacy outcome is the comparison of the incidence of complete healing of the target ulcer between the two treatment groups at the end of treatment.
  For the purpose of this study a complete healing will be defined as complete epithelialization which is maintained with no drainage for at least 2 weeks and is confirmed by a blinded assessor.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ON101 Cream | Aquacel® Hydrofiber® Dressing
Number analyzed (Participants) | 122 | 114
Participants | 74 | 40

2. Secondary Outcome: The Time of Healing Rate
Description: Time to complete ulcer healing, The time of the original healing will be taken as the time to healing.
Time Frame: 16 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | ON101 Cream | Aquacel® Hydrofiber® Dressing
Number analyzed (Participants) | 122 | 114
weeks | 14 [14.0 to 14.3] | NA [NA to NA] — unable to be estimated by Kaplan-Meier method due to some subjects are not completely healed

3. Secondary Outcome: Change in Ulcer Area
Description: Percentage change in ulcer surface area from baseline
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage change in ulcer surface area
Arm/Group | ON101 Cream | Aquacel® Hydrofiber® Dressing
Number analyzed (Participants) | 122 | 114
percentage change in ulcer surface area
  week 16 | -78 (42.6) | -78 (34.9)
  week 2 | -36 (32.9) | -38 (29.3)

4. Secondary Outcome: Percentage of Participants With a 50% Reduction of Ulcer Surface Area
Description: Percentage of subjects with a 50% reduction of ulcer surface area
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ON101 Cream | Aquacel® Hydrofiber® Dressing
Number analyzed (Participants) | 122 | 114
Participants | 101 | 98

5. Secondary Outcome: Incidence of Infection of the Target Ulcer
Description: Incidence of infection of the target ulcer
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ON101 Cream | Aquacel® Hydrofiber® Dressing
Number analyzed (Participants) | 122 | 114
Participants | 6 | 7

ADVERSE EVENTS:
Time Frame: Adverse event collection began after study intervention was initiated and continued through the entire study visit. (Day 1 to Day 197)
Arm/Group | ON101 Cream | Aquacel® Hydrofiber® Dressing
All-Cause Mortality (participants affected / at risk) | 1/122 | 0/114
Serious Adverse Events (participants affected / at risk) | 14/122 | 9/114
Other Adverse Events (participants affected / at risk) | 7/122 | 5/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ON101 Cream (N=122) | Aquacel® Hydrofiber® Dressing (N=114)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 2 (2)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ON101 Cream (N=122) | Aquacel® Hydrofiber® Dressing (N=114)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight increased (Investigations) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-25): https://cdn.clinicaltrials.gov/large-docs/23/NCT01898923/Prot_SAP_000.pdf